CLINICAL TRIAL: NCT03911336
Title: Harnessing Chronomodulation to Enhance Osteogenesis - A Pilot Randomized Controlled Trial -
Brief Title: Harnessing Chronomodulation to Enhance Osteogenesis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Decided not to proceed
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Satheesh Elangovan, Principal Investigator, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201904762
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Tooth Loss
Keywords: Chronotherapy; Chronomodulation; Osteogenesis; NSAID
MeSH Terms: conditions — Tooth Loss | interventions — Ketoprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: This study is designed as a parallel-arm, double-blinded pilot randomized controlled trial (RCT).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, Surgeon and Assessors collecting the data and conducting the appropriate statistical analyses for all outcomes in the study will be blinded.
  All surgical procedures will be scheduled between 8 and 10 AM and performed by the same blinded clinician to maintain a consistent therapeutic approach for all subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A - test (Experimental): Group A (Test) - Tooth extraction and intake of an NSAID (i.e. Ketoprofen ER 50 mg) at 8 AM and a non-NSAID (i.e. Acetaminophen / Paracetamol 500 mg) at 2 PM and 8 PM for a 3-day period, starting the regime at 2 PM on the day of the extraction.
  Interventions: Drug: Group A - test:Tooth extraction and intake of NSAID and a non-NSAID
- Group B - Control 1 (Active Comparator): Group B (Control 1) - Tooth extraction and intake of an NSAID (i.e. Ketoprofen ER 50 mg) at 8 PM and a non-NSAID (i.e. Acetaminophen / Paracetamol 500 mg) at 8 AM and 2 PM for a 3- day period, starting the regime at 2 PM on the day of the extraction.
  Interventions: Drug: Group B - Control 1: tooth extraction and intake of NSAID and a non-NSAID
- Group C - Control 2 (Active Comparator): Group C (Control 2) - Tooth extraction and intake of a non-NSAID (i.e. Acetaminophen / Paracetamol 500 mg) at 8AM, 2 PM and 8 PM for a 3-day period, starting the regime at 2 PM on the day of the extraction.
  Interventions: Drug: Group C - Control 2: tooth extraction and intake of a Non-Nsaid

INTERVENTIONS:
Drug: Group A - test:Tooth extraction and intake of NSAID and a non-NSAID — Tooth extraction and intake of an NSAID (i.e. Ketoprofen ER 50 mg) at 8 AM and a non-NSAID (i.e. Acetaminophen / Paracetamol 500 mg) at 2 PM and 8 PM for a 3-day period, starting the regime at 2 PM on the day of the extraction.
  Other Names: Ketoprofen ER 50 mg and Acetaminophen/Paracetamol 500 mg
  Arms: Group A - test
Drug: Group B - Control 1: tooth extraction and intake of NSAID and a non-NSAID — Tooth extraction and intake of an NSAID (i.e. Ketoprofen ER 50 mg) at 8 PM and a non-NSAID (i.e. Acetaminophen / Paracetamol 500 mg) at 8 AM and 2 PM for a 3-day period, starting the regime at 2 PM on the day of the extraction.
  Other Names: Acetaminophen/Paracetamol 500 mg and Ketoprofen ER 50 mg
  Arms: Group B - Control 1
Drug: Group C - Control 2: tooth extraction and intake of a Non-Nsaid — Tooth extraction and intake of a non-NSAID (i.e. Acetaminophen / Paracetamol 500 mg) at 8AM, 2 PM and 8 PM for a 3-day period, starting the regime at 2 PM on the day of the extraction.
  Other Names: Acetaminophen/Paracetamol 500 mg
  Arms: Group C - Control 2

SUMMARY:
Chronotherapy is an emerging field in biomedicine that leverages on fine-tuning the timing of drug delivery to obtain a therapeutic effect. Dr. Tamimi and his team have successfully harnessed chronotherapy using NSAIDs to enhance bone healing in a murine fracture model. Unpublished findings revealed that mice receiving carprofen for 3 days post-fracture exclusively during activity hours exhibited superior bone healing outcomes in comparison to specimens that received the same drug during resting hours.

This is a 3-arm RCT aimed at evaluating the effect of different chronotherapeutic NSAID regimens on intraoral bone healing in humans using an extraction socket healing model in the context of an early implant placement protocol.

The primary aim is to elucidate whether there are differences in osteogenesis and in the characteristics of the newly formed bone between patients following different post-operative NSAID chronotherapeutic protocols. Secondary endpoints of interest include assessment of alveolar bone and soft tissue dimensional changes between pre- and post-extraction, implant insertion torque, serum CRP levels, wound healing index and patient-reported discomfort at different time points.

If proven beneficial, the proposed chronotherapeutic approach could be readily implemented in clinical practice as a standalone therapy or as a valuable complement to existing standard-of-care protocols, due to its simplicity, safety and cost-effectiveness.

DETAILED DESCRIPTION:
Enrolled subjects will be randomly assigned to one of three groups (n=12 per group):

Group A (Test) - Tooth extraction and intake of an NSAID (i.e. Ketoprofen ER 50 mg) at 8 AM and a non-NSAID (i.e. Acetaminophen / Paracetamol 500 mg) at 2 PM and 8 PM for a 3-day period, starting at 2 PM on the day of the extraction.

Group B (Control 1) - Tooth extraction and intake of an NSAID (i.e. Ketoprofen ER 50 mg) at 8 PM and a non-NSAID (i.e. Acetaminophen / Paracetamol 500 mg) at 8 AM and 2 PM for a 3-day period, starting at 2 PM on the day of the extraction.

Group C (Control 2) - Tooth extraction and intake of a non-NSAID (i.e. Acetaminophen / Paracetamol 500 mg) at 8AM, 2 PM and 8 PM for a 3-day period, starting at 2 PM on the day of the extraction.

VISIT 1 - Screening Referred or self-referred subjects that appear to meet all the eligibility criteria upon phone pre-screening will be invited to an in-person screening visit at the UICOD. The study purpose, duration, potential risks and expected benefits will be explained in detail to the subjects, as part of the consenting process. All screened subjects will be provided with hard copies of the study timeline and the signed consent form. Upon medical and dental history review, as well as site-specific clinical and radiographic evaluation, eligible subjects interested in participating in the study will be scheduled for Visit 2. Intraoral photographs of the site of interest will be taken. Additionally, a cone-beam computed tomography (CBCT) scan will be obtained and interpreted to evaluate the study site, prior to the baseline intervention.

VISIT 2 - Tooth Extraction (Baseline Intervention) Medical and dental history will be reviewed and updated, if necessary. Subsequently, subjects will be asked to sign the surgical procedure consent form. Prior to tooth extraction, an intraoral scan of the area of interest will be obtained using a digital scanner (e.g. Planmeca Emerald S). Likewise, a blood sample (~ 4.5 cc) will be collected for serum C-reactive protein (CRP) analysis. Following administration of local infiltrative anesthesia, the study tooth will be extracted in a minimally traumatic fashion, avoiding flap reflection. Following tooth extraction, the socket walls will be carefully inspected for the existence of dehiscences or fenestrations. Sites presenting a bony defect affecting >20% of the total wall height will be excluded. Site will be sealed using a collagen matrix (Mucograft Seal, Geistlich Pharma) stabilized with simple interrupted sutures. The intervention will be documented using intraoral photography.

Upon completion of the intervention, subjects will be randomly assigned to one of the study groups and provided with detailed written and verbal post-operative instructions, including a drug diary specific to the group that they are allocated in and a visual analog scale (VAS) to record their perceived discomfort at day 0, 1, 2, 3 and 7 after the intervention.

VISIT 3 - Postoperative Evaluation Any medical or dental history changes, or adverse events will be recorded. Sutures will be removed. An intraoral scan and photographs of the site will be obtained. Visual assessment of the healing status will be made using a wound healing index (WHI). Biofilm on the adjacent teeth will be removed and home care instructions will be revisited.

VISIT 4 - Implant Placement At the beginning of this visit, a second segmental CBCT scan will be obtained, using the same settings employed at baseline. CBCT images will be employed to evaluate ridge dimensional changes compared to baseline, as well as bone availability for dental implant placement. Any medical or dental history changes, or adverse events will be recorded. A blood sample (~ 4.5 cc) and an intraoral scan will be obtained. Assessment of the healing status will be made using the aforementioned WHI. After administering local infiltrative anesthesia, patients will undergo implant insertion, according to the early implant placement protocol.10 Following full-thickness flap elevation, a bone core biopsy of the study site will be obtained using a trephine drill of 2.5 mm in diameter or wider. The bone core will be immediately submerged in a solution of 10% neutral buffered formalin (NBF) for microCT (µCT) and histological analyses.

Implant site preparation and placement will be conducted according to the manufacturer's recommendations (SLActive Bone Level - Straumann AG). Implant insertion torque will be recorded. Intraoral periapical radiographs will be obtained, as necessary, in order to assess implant placement location. Following final implant placement and cover screw delivery, simultaneous buccal contour augmentation will be performed via guided bone regeneration (GBR) using a dual bone graft. This graft composite will consist of an initial layer of locally harvested autogenous bone to cover the exposed implant surface, combined with a superficial layer of deproteinized bovine bone particles (DBBM; BioOss granules 0.25 - 1.0 mm, Geistlich Pharma), which will be subsequently covered with a native porcine collagen membrane (Bio-Gide; Geistlich Pharma). All procedures will be executed according to a two-stage (submerged) approach. Therefore, tension-free primary soft tissue closure will be attained. The procedure will be documented with intraoral photographs. All subjects will be provided with detailed written and verbal post-operative instructions. They will be instructed to avoid any disturbance in the surgical area for two weeks. Patients will be asked to use a mouthwash containing 0.12% of chlorhexidine gluconate twice a day, thirty seconds at a time, avoiding any eating or drinking for 30 minutes after rinsing, starting 48 hours after the baseline intervention. Post-operative medications (e.g. antibiotics, anti-inflammatory drugs and analgesics) will be prescribed on an individual basis.

VISIT 5 - Postoperative Evaluation (Final Study Visit) This visit will be scheduled at approximately two weeks after implant placement. Any medical or dental history changes, or adverse events will be recorded. Intraoral photographs of the site of interest, will be obtained. Assessment of the healing status will be made using the aforementioned WHI. All remaining sutures will be removed. Biofilm on the adjacent teeth will be removed and home care instructions will be revisited. Upon completion of this final study visit, the patient will be entered in a regular patient care routine, including scheduling of a future visit for implant uncovering in no less than 4 months and later referral to the restorative dentist, in order to complete tooth replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older) males or females with an ASA status of I or II and adequate physical and mental health to undergo study-related procedures
* In need of extraction of a maxillary incisor, maxillary or mandibular canine, or maxillary or mandibular premolar and successive tooth replacement therapy according an early implant placement protocol10
* Extractions socket walls must be intact or have no more than one bony wall dehiscence or fenestration extending no more than 20% of the total bony wall height
* Subjects must have read, understood and signed the informed consent form

Exclusion Criteria:

* Acute infection associated with the tooth to be extracted or with adjacent teeth
* Known allergies or medical contraindications to any of the study-related drugs and biologic materials
* Sleeping disorders or jet lagged from a recent trip or working in night shift jobs
* History of significant heart, stomach, liver, kidney, blood, immune system disease, or other organ impairment or systemic diseases or disorders that may prevent undergoing the proposed treatment and/or may significantly affect bone healing (e.g. uncontrolled diabetes, thyroid disorders or Paget's disease)
* Current smokers or former smokers who quit less than 12 months prior to the initiation of the study
* Subjects taking any medication or supplement known to influence bone metabolism, such as IV bisphosphonates, long-term history of oral bisphosphonates or chronic intake of glucocorticoids
* Regular or within 7 days of baseline intake of any anti-inflammatory and/or analgesic drugs
* Need of oral or intravenous sedation
* Pregnant women or nursing mothers
* History of recreational drug abuse and/or heavy alcohol use
* History of lack of compliance with dental visits or unwilling to return for the required number of visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
proportion (%) of mineralized tissue | 6 weeks after extraction
  proportion (%) of mineralized tissue present in the bone core samples obtained at the time of implant placement, approximately 6 weeks after tooth extraction. This will be evaluated via histomorphometric analysis.

SECONDARY OUTCOMES:
µCT analysis | 6 weeks post-extraction
  Characteristics of mineralized tissue evaluated via μCT analysis.
Alveolar bone variations | Baseline to 6 weeks post-extraction
  Bone linear and volumetric dimensional changes between visits 2 and 4 via DICOM data analysis.
Alveolar ridge contour variations | Baseline to 6 weeks post-extraction
  Alveolar ridge contour variations from visits 2 to visit 5 via STL data analysis.
Implant insertion torque | 6 weeks post-extraction
  Implant insertion torque at visit 4, expressed in N/cm
Serum CRP | Baseline
  Serum CRP assessment using circulating blood samples obtained at visits 2 and 4
Serum CRP | 6 weeks post-extraction
  Serum CRP assessment using circulating blood samples obtained at visits 2 and 4
Wound Healing Index (WHI) | 1 week post-extraction
  WHI assessment at visit 3
Wound Healing Index (WHI) | 6 weeks post-extraction
  WHI assessment at visit 4
Wound Healing Index (WHI) | 8 weeks post-extraction
  WHI assessment at visit 5
Patient Reported Outcome Measures (PROMS) | Baseline
  Self-perceived discomfort measured using a 10-point Visual Analog Scale (1 [lower discomfort] to 10 [higher discomfort]) at day 0, 1, 2, 3 and 7 after tooth extraction
Patient Reported Outcome Measures (PROMS) | Day 1 post-extraction
  Self-perceived discomfort measured using a 10-point Visual Analog Scale (1 [lower discomfort] to 10 [higher discomfort]) at day 0, 1, 2, 3 and 7 after tooth extraction
Patient Reported Outcome Measures (PROMS) | Day 2 post-extraction
  Self-perceived discomfort measured using a 10-point Visual Analog Scale (1 [lower discomfort] to 10 [higher discomfort]) at day 0, 1, 2, 3 and 7 after tooth extraction
Patient Reported Outcome Measures (PROMS) | Day 3 post-extraction
  Self-perceived discomfort measured using a 10-point Visual Analog Scale (1 [lower discomfort] to 10 [higher discomfort]) at day 0, 1, 2, 3 and 7 after tooth extraction
Patient Reported Outcome Measures (PROMS) | Day 7 post-extraction
  Self-perceived discomfort measured using a 10-point Visual Analog Scale (1 [lower discomfort] to 10 [higher discomfort]) at day 0, 1, 2, 3 and 7 after tooth extraction

CONTACTS AND LOCATIONS:
Overall Officials: Satheesh Elangovan, BDS DSc DMSc, Study Chair — University of Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slade GD, Akinkugbe AA, Sanders AE. Projections of U.S. Edentulism prevalence following 5 decades of decline. J Dent Res. 2014 Oct;93(10):959-65. doi: 10.1177/0022034514546165. Epub 2014 Aug 21. PMID 25146182
- [Background] Elani HW, Starr JR, Da Silva JD, Gallucci GO. Trends in Dental Implant Use in the U.S., 1999-2016, and Projections to 2026. J Dent Res. 2018 Dec;97(13):1424-1430. doi: 10.1177/0022034518792567. Epub 2018 Aug 3. PMID 30075090
- [Background] Innominato PF, Roche VP, Palesh OG, Ulusakarya A, Spiegel D, Levi FA. The circadian timing system in clinical oncology. Ann Med. 2014 Jun;46(4):191-207. doi: 10.3109/07853890.2014.916990. PMID 24915535
- [Background] Takahashi JS, Hong HK, Ko CH, McDearmon EL. The genetics of mammalian circadian order and disorder: implications for physiology and disease. Nat Rev Genet. 2008 Oct;9(10):764-75. doi: 10.1038/nrg2430. PMID 18802415
- [Background] Giacchetti S, Bjarnason G, Garufi C, Genet D, Iacobelli S, Tampellini M, Smaaland R, Focan C, Coudert B, Humblet Y, Canon JL, Adenis A, Lo Re G, Carvalho C, Schueller J, Anciaux N, Lentz MA, Baron B, Gorlia T, Levi F; European Organisation for Research and Treatment of Cancer Chronotherapy Group. Phase III trial comparing 4-day chronomodulated therapy versus 2-day conventional delivery of fluorouracil, leucovorin, and oxaliplatin as first-line chemotherapy of metastatic colorectal cancer: the European Organisation for Research and Treatment of Cancer Chronotherapy Group. J Clin Oncol. 2006 Aug 1;24(22):3562-9. doi: 10.1200/JCO.2006.06.1440. PMID 16877722
- [Background] Cutolo M. Glucocorticoids and chronotherapy in rheumatoid arthritis. RMD Open. 2016 Mar 18;2(1):e000203. doi: 10.1136/rmdopen-2015-000203. eCollection 2016. PMID 27042335
- [Background] Okazaki F, Matsunaga N, Hamamura K, Suzuki K, Nakao T, Okazaki H, Kutsukake M, Fukumori S, Tsuji Y, To H. Administering xCT Inhibitors Based on Circadian Clock Improves Antitumor Effects. Cancer Res. 2017 Dec 1;77(23):6603-6613. doi: 10.1158/0008-5472.CAN-17-0720. Epub 2017 Oct 16. PMID 29038345
- [Background] Swanson CM, Kohrt WM, Buxton OM, Everson CA, Wright KP Jr, Orwoll ES, Shea SA. The importance of the circadian system & sleep for bone health. Metabolism. 2018 Jul;84:28-43. doi: 10.1016/j.metabol.2017.12.002. Epub 2017 Dec 9. PMID 29229227
- [Background] Dallmann R, Okyar A, Levi F. Dosing-Time Makes the Poison: Circadian Regulation and Pharmacotherapy. Trends Mol Med. 2016 May;22(5):430-445. doi: 10.1016/j.molmed.2016.03.004. Epub 2016 Apr 5. PMID 27066876
- [Background] Chappuis V, Rahman L, Buser R, Janner SFM, Belser UC, Buser D. Effectiveness of Contour Augmentation with Guided Bone Regeneration: 10-Year Results. J Dent Res. 2018 Mar;97(3):266-274. doi: 10.1177/0022034517737755. Epub 2017 Oct 26. PMID 29073362